CLINICAL TRIAL: NCT04767555
Title: Impact of ILM Peeling on Functional and Anatomic Outcomes of Vitrectomy for Primary Rhegmatogenous Retinal Detachment - the I-Peel Study
Brief Title: Impact of ILM Peeling in RRD/ I-Peel
Acronym: I-Peel
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berner Augenklinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-Peel 2021-00027
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Retinal Detachment
Keywords: retinal detachment; ILM-peeling
MeSH Terms: conditions — Retinal Detachment | interventions — Tooth Exfoliation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ILM (inner limiting membrane) peeling (Experimental): ILM peeling adding to standard vitreous surgery in patients suffering from retinal detachment
  Interventions: Procedure: ILM (inner limiting membrane) peeling
- No Peeling (No Intervention): standard vitreous surgery without ILM peeling in patients suffering from retinal detachment

INTERVENTIONS:
Procedure: ILM (inner limiting membrane) peeling — The standard technique for the removal of the inner limiting membrane is a dye-assisted ILM peeling established since 20 years as the standard of care to treat vision loss due to epiretinal membranes or macular holes in eyes with an otherwise stable retina, but not during retinal detachment surgery. Other dyes may show a stronger staining effect but since there is evidence of a potential toxicity of ICG the investigators use the well-tolerated and for this purpose approved trypan blue dye Membrane Blue ® (Dorc). This intervention will be performed in addition to standard vitreoretinal re-attachment surgery.
  Arms: ILM (inner limiting membrane) peeling

SUMMARY:
Retinal detachment is associated with a substantial risk of re-detachment in 10-20% and to the formation of secondary epiretinal membranes in up to 15%. Relevant postoperative vision loss is encountered in many instances, primarily in consequence of macular involvement, but also secondarily due to postoperative complications, namely the formation of an epiretinal membrane and proliferative vitreoretinopathy. These mechanical reasons of influence can potentially be prevented by ILM peeling during reattachment surgery. This, however, is not a generally accepted standard of care during primary routine vitrectomy.

Two groups suffering from primary retinal detachment will be compared: the first group will receive standard re-attachment vitrectomy surgery, whereas the second group will receive an identical vitrectomy surgery, but with additional ILM peeling. In this study, the investigators wish to assess the influence of ILM peeling on visual outcomes and postoperative complications over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* primary rhegmatogenous retinal detachment
* of legal age (18 years or older)
* in case of bilateral retinal detachment, only the first-affected eye will be included

Exclusion Criteria:

* pre-existing functional and morphological changes to the macula, hindering visual recovery (amblyopia, trauma, macular degeneration)
* advanced retinal detachment with PVR stage C2 or more
* eyes pre-operated within six months prior to the development of RD
* state after any vitreoretinal surgery
* state after complicated cataract surgery, including aphakia and anterior chamber lens implantation
* patients with increased risk profiles
* myopia magna (≥7 diopters)
* advanced diabetic retinopathy
* any chronic ocular or systemic inflammatory disease
* any other proliferative systemic disease or condition associated with impaired wound healing

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients developing secondary epiretinal membrane formation | 12 months
  Clinically significant secondary epiretinal membrane formation requiring revision surgery

SECONDARY OUTCOMES:
Rate of re-detachments in patients | 12 months
  Revision surgery due to re-detachment independently of secondary epiretinal membrane formation
Best-corrected visual acuity | 12 months
  Change in best-corrected visual acuity
Complication rates | 12 months
  Intra- and postoperative complication rates including PVR
Surgical times | minutes (0-300)
  How long does the surgery take

CONTACTS AND LOCATIONS:
Overall Officials: Justus G Garweg, Prof. Dr., Principal Investigator — Berner Augenklinik
Locations (1):
- Berner Augenklinik, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aras C, Arici C, Akar S, Muftuoglu G, Yolar M, Arvas S, Baserer T, Koyluoglu N. Peeling of internal limiting membrane during vitrectomy for complicated retinal detachment prevents epimacular membrane formation. Graefes Arch Clin Exp Ophthalmol. 2009 May;247(5):619-23. doi: 10.1007/s00417-008-1025-y. Epub 2008 Dec 24. PMID 19107502
- [Background] Garweg JG, Bergstein D, Windisch B, Koerner F, Halberstadt M. Recovery of visual field and acuity after removal of epiretinal and inner limiting membranes. Br J Ophthalmol. 2008 Feb;92(2):220-4. doi: 10.1136/bjo.2007.131862. Epub 2007 Nov 30. PMID 18055572
- [Background] Garweg JG, Deiss M, Pfister IB, Gerhardt C. IMPACT OF INNER LIMITING MEMBRANE PEELING ON VISUAL RECOVERY AFTER VITRECTOMY FOR PRIMARY RHEGMATOGENOUS RETINAL DETACHMENT INVOLVING THE FOVEA. Retina. 2019 May;39(5):853-859. doi: 10.1097/IAE.0000000000002046. PMID 29394235
- [Background] Hohn F, Kretz FT, Pavlidis M. [Primary vitrectomy with peeling of the internal limiting membrane under decaline: a promising surgical maneuver for treatment of total and subtotal retinal detachment]. Ophthalmologe. 2014 Sep;111(9):882-6. doi: 10.1007/s00347-014-3158-1. German. PMID 25204530
- [Background] Kodjikian L, Richter T, Halberstadt M, Beby F, Flueckiger F, Boehnke M, Garweg JG. Toxic effects of indocyanine green, infracyanine green, and trypan blue on the human retinal pigmented epithelium. Graefes Arch Clin Exp Ophthalmol. 2005 Sep;243(9):917-25. doi: 10.1007/s00417-004-1121-6. Epub 2005 Apr 15. PMID 15834606
- [Background] Koerner F, Garweg J. Advances in the management of vitreomacular traction syndrome and macular hole. Dev Ophthalmol. 1997;29:15-29. doi: 10.1159/000060723. No abstract available. PMID 9413690
- [Background] Odrobina D, Bednarski M, Cisiecki S, Michalewska Z, Kuhn F, Nawrocki J. Internal limiting membrane peeling as prophylaxis of macular pucker formation in eyes undergoing retinectomy for severe proliferative vitreoretinopathy. Retina. 2012 Feb;32(2):226-31. doi: 10.1097/IAE.0b013e31821a12e9. PMID 21878849